CLINICAL TRIAL: NCT06288347
Title: A Cross-over Randomized-control Study Evaluating the Efficacy of GGON in Reducing Maladaptive Beliefs Related to Orthorexia Nervosa.
Brief Title: Study of the Efficacy of GGON: a Cognitive Training App for Orthorexia Nervosa.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María Roncero, Associate Professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 216099
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Orthorexia Nervosa
Keywords: maladaptive beliefs; cognitive therapy; mobile app; e-health
MeSH Terms: conditions — Orthorexia Nervosa

STUDY DESIGN:
Intervention Model Description: All participants were requested to complete web-based assessment, with questionnaires relating to maladaptive beliefs associated with ON, ortorexia, eating and depressive symptomatology, obsessive belifs and self-esteem at baseline (T1).
  The experimental group started using the app for 15 days, and later completed the following assessment (T2). The control group also completed the T2 in the same date but started to use the app after this second assessment.15 days and one month later, both groups completed T3 and T4.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group used the GGON module for 15 days after the first assessment.
  Interventions: Device: GGON mobile app.
- Control group (Active Comparator): The control group used the GGON module for 15 days after the second assessment.
  Interventions: Device: GGON mobile app.

INTERVENTIONS:
Device: GGON mobile app. — The intervention will be done through an app named GGON, which is used to work on the dysfunctional beliefs that are associated with orthorexia nervosa. The app is made up of a series of levels comprising the topics based in cognitive-conductual perspective that are related to Orthorexia Nervosa. At each level, affirmations in the form of beliefs appear on the screen, and the person must accept them if they are functional, adaptive and positive; or reject them if they are dysfunctional, maladaptive and negative.

SUMMARY:
The aim of the present study is to evaluate the efficacy of GGON to decrease the maladaptive beliefs associated with orthorexia nervosa (ON) in non-clinical adult population. Specifically, a randomized controlled trial with crossover assignment design and two groups (experimental and control) will be carried out in adults aged 18-65 years to assess the changes pre and post use the app. It's expected that after the use of the GGON app for 15 days are, at the primary level: decrease in the degree of ascription to dysfunctional beliefs associated with ON; and at the secondary level: decrease in orthorexia nervosa symptomatology, in eating symptomatology and in obsessive beliefs; increase in self-esteem; and no changes in drepessive symptomatology. These results are also expected to be maintained in subsequent follow-ups, at 15 days and a month after to finish the app in experimental group, and 15 days after to finish the app in control group.

DETAILED DESCRIPTION:
There is a digital platform called GGtude, which is composed of different modules, each of them aimed at working with different mental health problems. The goal is to provide an easy-to-use tool as a CBT complement to work on the self-dialogue that relates to the core beliefs associated with the psychological problem in particular. To achieve this target, a cognitive training exercise is performed: different sentences appear in the form of beliefs, and the person must identify and accept those beliefs that are functional, adaptive and positive, dragging them to the lower part of the screen; and reject those that are dysfunctional, maladaptive and negative dragging them to the upper part of the screen.

There are different modules, for example, to work self-esteem, eating disorders, depression, body image or obsessive-compulsive disorder, that have proven their effectiveness. The GGON app has not efficacy studies. So, it is relevant to evaluate its effectiveness with an RCT study.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65.
* Have a dispositive with Internet access.

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Change in the degree of ascription to dysfunctional beliefs associated with Orthorexia Nervosa | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in the degree of ascription to dysfunctional beliefs associated with Orthorexia Nervosa measured by Orthorexia Beliefs Scale (OBS). Self-assessment instrument that evaluates the core beliefs of orthorexia nervosa. Its original version is in Spanish. It is composed of 21 items with a 4-point Likert-type scale response (0 = Strongly Disagree to 3 = Strongly Agree). Specifically, it assesses three factors: value, morality and control. These factors present adequate internal consistency in the sample of this study, with Cronbach's α values ranging from .72 to .86.

SECONDARY OUTCOMES:
Change in Orthorexia symptomatology | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in Orthorexia symptomatology measured by Teruel Orthorexia Scale (TOS). It is an instrument for the assessment of orthorexia. Its original version is in Spanish. It consists of 17 items with a 4-point Likert-type response scale (0 = Strongly disagree to 3 = Strongly agree). It evaluates two factors: Healthy Orthorexia, referring to a healthy interest in diet, not associated with psychopathology; and Orthorexia Nervosa, which is the pathological preoccupation with a healthy diet. In the current study these factors present very good internal consistency, with Cronbach's α values of .84 and .82.
Change in eating symptomatology | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in eating symptoms measured by the Eating Disorder Examination Questionnaire (EDE-Q). It is a 36-item questionnaire designed to evaluate the range, frequency and severity of behaviors associated with eating disorders. It is structured into four distinct subscales: restriction, food concern, weight concern, and figure concern, each encompassing attitudinal and behavioral components. In the current study exclusively 22 attitudinal inquiries were used. Responses to these inquiries are assessed on a 7-point Likert scale, spanning from 0 ("No day/ No time/ Not at all") to 6 ("Every day/ Always/ Completely"). Internal consistency values for such factors were very good in this study (Cronbach's αs ranging from .81 to .92).
Change in self-esteem. | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in self-report measures with The Single-Item Self-Esteem Scale (SISE). It is a self-esteem questionnaire in which individuals are asked to rate the extent to which the statement "I have high self-esteem" matches their self-perception on a 9-point scale (ranging from 1 = "Not very true for me" to 9 = "Very true for me"). This scale demonstrates strong test-retest reliability and exhibits a criterion validity coefficient comparable to that of the Rosenberg Self-Esteem Scale (Rosenberg, 1965), exceeding .80 Cronbach's alpha value.
Change in emotional symptomatology | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in emotional symptomatology measured by The Depression, Anxiety-Stress Scale (DASS-21). It is a self-report that assesses negative emotional symptoms: depression, anxiety and stress. It consists of 21 items that are answered on a Likert-type scale from 0 to 3 (0 = "It does not affect me at all" and 4 = "It affects me a lot or most of the time"). In the present study, only the 7-itmes depression scale was used, which presented a very good internal consistency in this sample, with Cronbach's alpha values of .91.
Change in obsessive beliefs | 15 days, and for experimental group 15 and 30 days later; and for the control group 15 days later
  Score change in obsessive beliefs measured by Inventario de Creencias Obsesivas Revisado (ICO-R). It is a 50-items questionnaire which assesses the dysfunctional beliefs related to development or mantenaince of obsessive-compulssive disorder (OCD), in both clinical and non-clinical samples. Its original version is in Spanish. It has a 7-point Likert-type response scale from 1 "strongly disagree" to 7 "strongly agree". It evaluates 8 scales: excessive responsibility, importance of thought control, perfectionism, overestimation of danger, intolerance to uncertainty, overimportance of thoughts, thought-action probability fusion, and thought-action moral fusion. Only the 33 items corresponding to the factors of excessive responsibility, importance of thought control, perfectionism, overestimation of danger and intolerance to uncertainty were used in this study. These factors present very good internal consistency in this sample, with Cronbach's α values ranging from .79 to .89.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in a publication.
Time Frame: 3 months after the study is published.
Access Criteria: The variables analyzed will be included in the manuscript in which the RCT data are presented, and will be published on the institutional page of the applicants' university (https://roderic.uv.es/) up to 3 months after the article is published.
URL: http://roderic.uv.es

REFERENCES:
- See also: Description Information about GGTUDE Mobile App and links to download. — http://ggapps.net/2018/04/11/ggro-relationship-obsession-rocd/

DOCUMENTS (1):
  • Informed Consent Form (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT06288347/ICF_000.pdf